CLINICAL TRIAL: NCT03498001
Title: Effects of GLP-1 Agonists on CArdiac Steatosis Evaluated by Magnetic Resonance Imaging
Acronym: LICAS-MR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUENANCIA APJ 2016
Record Dates: First submitted 2018-03-30; First posted 2018-04-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucagon-Like Peptide-1 Receptor Agonists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Drug: GLP-1 agonists; Procedure: Cardiac MRI; Other: Follow up by phone

INTERVENTIONS:
Drug: GLP-1 agonists — Liraglutide: 6 mg/ml Semaglutide: 1.34 mg/ml Dulaglutide: de 0.75 mg ou 1.5 mg
Procedure: Cardiac MRI — T3 myocardial MRI (total acquisition time : 1h) performed before initiation of treatment and measuring the concentration of intramyocardial triglycerides ([TG] by NMR spectroscopy, parameters of cardiac morphology (myocardial mass, (epicardial fat surface, pericardial fat surface), function (LVEF, SV, TDV, PFR, TPFR) and tissue parameters (extracellular volume, left myocardial fibrosis volume).
Other: Follow up by phone — at 2 and 4 mois

SUMMARY:
Type II diabetes is a known risk factor for heart failure, particularly through the progressive development of diabetic cardiomyopathy. Cardiac metabolic parameters, including myocardial steatosis and epicardial fat, are altered in diabetic patients. The development of new anti-diabetics (incretins) has demonstrated protective cardiovascular effects independent of effects on glycemic control for the first time in the history of these therapies. Thus Glucagon-Like Peptide 1 (GLP-1) agonists improve the recovery of cardiac function after a heart attack and decrease atheromatous processes. It has also been demonstrated in a diabetic rat model that the administration of Liraglutide, a GLP-1 agonist, leads to normalization of myocardial steatosis associated with beneficial cardiac molecular remodeling involving pro-apoptotic, oxidative and metabolic processes. These beneficial cardiovascular effects were observed in the absence of any changes in blood glucose, insulin levels or body weight.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has given his consent
* Adult patient over 50 years of age Type II diabetic treated without modification of the antidiabetic treatment during the previous 3 months
* HbA1c ≥ 7%.
* Patient for whom a decision to start a GLP-1 agonist treatment has been made (Liraglutide, Semaglutide, Dulaglutide).
* At least one risk factor from among:
* Treated hypertension,
* treated dyslipidemia,
* History of obesity (BMI>30 kg/m2)
* Active smoking (from 1 cigarette per day) or smoking cessation for less than 3 years,
* Coronary heredity (myocardial infarction or sudden death before age 55 in father/brother, myocardial infarction or sudden death before age 65 in mother/sister)

Exclusion Criteria:

- Protected adult Patient not affiliated to a national health insurance scheme Pregnant or breastfeeding woman Women who intend to become pregnant or of childbearing age and do not use adequate contraceptive methods.

Antidiabetic treatment of the incretin family (DPP4 inhibitor except sitagliptin) Severe renal failure (clearance <30ml/min according to Cockroft due to gadolinium injection) Claustrophobia / contraindication to MRI (compatible non-MRI implanted metallic material) History of hypersensitivity to gadoteric acid or gadolinium-based contrast agents and meglumine Hypersensitivity to Liraglutide, Semaglutide, Dulaglutide or any of the excipients History or presence of pancreatitis (acute or chronic) Chronic inflammatory bowel disease Diabetic gastroparesis Dysthyroidism

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Concentration of intramyocardial triglycerides at 6 months | Month 6
  Intramyocardial triglyceride concentration, expressed in %, evaluated by NMR spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Houbachi L, Walker PM, Fournel I, Ksiazek E, Petit JM, Cochet A, Leclercq T, Roger A, Simoneau I, Bouillet B, Guenancia C. Evolution of myocardial steatosis in high cardiovascular risk T2DM patients treated by GLP1 receptor agonists: LICAS study. Diabetes Res Clin Pract. 2025 Mar;221:112017. doi: 10.1016/j.diabres.2025.112017. Epub 2025 Feb 1. PMID 39900263